CLINICAL TRIAL: NCT00553566
Title: Bladder Cancer Prognosis Programme (Incorporating SELENIB Trial) [COHORT]
Brief Title: Effect of Dietary, Lifestyle, and Environmental Factors on Patients With Early-Stage Bladder Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Birmingham (Other)
Organization: National Cancer Institute (NCI) (NIH)
Other Study IDs: CDR0000574078; CRUK-BCPP-2005-01-COHORT; ISRCTN13889738; EU-20768
Record Dates: First submitted 2007-11-02; First posted 2007-11-05 (Estimated); Last update posted 2014-01-10 (Estimated); Status verified 2010-02

CONDITIONS: Bladder Cancer
Keywords: stage 0 bladder cancer; stage I bladder cancer; transitional cell carcinoma of the bladder
MeSH Terms: conditions — Urinary Bladder Neoplasms

INTERVENTIONS:
Procedure: medical chart review
Procedure: questionnaire administration
Procedure: study of socioeconomic and demographic variables

SUMMARY:
RATIONALE: Learning about the long-term effects of dietary, lifestyle, and environmental factors on the risk of cancer progression and recurrence may help the study of bladder cancer in the future.

PURPOSE: This clinical trial is studying how dietary, lifestyle, and environmental factors affect patients with early-stage bladder cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To examine if common and potentially modifiable dietary, lifestyle, and environmental exposures affect the risk of recurrence and progression in bladder cancer.

OUTLINE: This is a multicenter study.

Detailed information will be collected about the patients' lifestyle and their exposure to risk factors associated with bladder cancer using semi-structured questionnaires. A baseline questionnaire will be administered at the time of diagnosis and will collect information about socio-demographics, environmental exposures, medical history, diet, health-related quality of life, and social support.

Further questionnaires will be administered at regular follow-up visits to capture information relating to changes in exposure. A postal questionnaire will be used to collect historical information that may require the patient to check records or consult family or friends. Patients will also be asked to keep a 1-week food, fluid, and micturition diary.

Patients continue to complete questionnaires at 3 months and then annually for up to 5 years.

Peer Reviewed and Funded or Endorsed by Cancer Research UK.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

Inclusion criteria:

* Enrolled on parent protocol CRUK-BCPP-2005-01
* Bladder lesion with cystoscopic characteristics compatible with urothelial cancer or transitional cell carcinoma
* Histologically proven urothelial cancer meeting one of the following criteria:

  * Stage Ta (WHO grade 2/3, or grade 1 tumors that are either multifocal or > 3 cm in size)
  * Stage T1 (any grade)
  * Stage Tis

Exclusion criteria:

* Previous diagnosis of cancer of the urethra, bladder, ureter, or renal pelvis within the 10 years prior to current diagnosis

PATIENT CHARACTERISTICS:

Inclusion criteria:

* Fit for cystoscopy and surgical biopsy/resection

Exclusion criteria:

* HIV infection
* Any condition that, in the opinion of the local investigator, might interfere with the safety of the patient or evaluation of the study objectives

PRIOR CONCURRENT THERAPY:

* Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1600
Dates: Start 2005-12

PRIMARY OUTCOMES:
Recurrence at 5 years
Progression at 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Maurice Zeegers, Study Chair — University of Birmingham
Locations (1):
- University of Birmingham, Edgbaston, England, United Kingdom